CLINICAL TRIAL: NCT04260373
Title: A Phase I Mass Balance and Biotransformation Study of [14C]SHR4640 in Chinese Healthy Adult Male Volunteers.
Brief Title: Study to Evaluate the Mass Balance and Biotransformation of [14C]SHR4640 in Chinese Healthy Adult Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHR4640-106
Record Dates: First submitted 2020-01-20; First posted 2020-02-07 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Healthy Adult Male Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]SHR4640 (Experimental): Patients will receive single dose of [14C]SHR4640 (Suspension, 10mg/80μCi).
  Interventions: Drug: [14C]SHR4640

INTERVENTIONS:
Drug: [14C]SHR4640 — Patients will receive single dose of orally [14C]SHR4640 on Day 1.

SUMMARY:
Study to Evaluate the Mass Balance and Biotransformation of Single Dose [14C]SHR4640 in Chinese healthy adult male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Signing the informed consent forms;
2. Healthy adult males;
3. Age: 18 Years to 45 Years(Including the boundary value);
4. Weight: Body mass index(BMI) between 19 and 26 kg/m2(Including the boundary value);

Exclusion Criteria:

1. Persons with abnormal physical examination, routine laboratory examination (blood routine, urine routine, stool routine + occult blood, blood biochemistry, blood coagulation routine, thyroid function), complete set of sex hormones, 12-lead electrocardiogram, X-ray (orthotopic), abdominal b-ultrasound (liver, bile, pancreas, spleen and kidney) and clinical significance;
2. Hepatitis b surface antigen, e antigen, hepatitis c antibody, HIV antibody and syphilis antibody, any one of these is positive.
3. Any medication taken within 14 days prior to screening;
4. Taking any clinical trial drug or participating in any clinical trial of any drug within 3 months prior to the screening period or preparing to participate in any other clinical trial within 1 month after the end of this trial;
5. Persons with history of organic heart disease, heart failure, myocardial infarction, angina pectoris, cardiac arrhythmias can not be explained, reverse sexual ventricular tachycardia, ventricular tachycardia, lengthened QT syndrome history or have QT syndrome symptoms and family history;
6. Persons who underwent major surgery within 6 months before the screening period or the surgical incision was not completely healed;Major surgery includes, but is not limited to, any operation with significant risk of bleeding, prolonged general anesthesia, open biopsy or significant traumatic injury;
7. A history of any clinical serious illness or disease or condition that the investigator believes may affect the results of the study, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary or blood, immune, mental and metabolic diseases;
8. Subject with known hypersensitivity or allergy to SHR4640, or any component of SHR4640;
9. Hemorrhoids or perianal disease with regular/ongoing hematochezia;
10. Subjects who have habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease;
11. Those who have history of alcohol abuse 1 month prior to screening period, or the alcohol breath test results ≥20 mg/dl during screening period；
12. Subjects who smoked daily >5 sticks of cigarette 3 months prior to first dose or cannot give up smoking during study;
13. Subjects who have history of drug abuse or taking soft drug (i.e., marihuana) 3 months prior to screening period or taking hard drugs (i.e., cocaine, amphetamines, benzodiazepine, etc.); or the results of urine test in drugs were positive;
14. Subjects who were used to drink grapefruit juice or overconsumption of tea, coffee, and the drink with caffeine; and cannot give up them during test;
15. Subjects who need long-term exposure to radiation, or who have been exposed to PET-CT or ECT within 3 months prior to study drug administration or who have participated in the labeling test of radiopharmaceuticals;
16. Subjects who have fertility planning within the range of starting trial - 1 year after finishing trial;
17. Subjects who have excessive bleeding or blood donation (400ml) 3 months prior to screening period, or planned to donate blood 1 month after finishing this trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Quantitive analysis of whole radioactivity of excrement of orally administered [14C]SHR4640 in Chinese healthy adult male volunteers to obtain the mass balance data and the main excretion pathway in human body by liquid scintillation counter. | Up to 10 days (approx) from the start of administration.
  The percentage of radioactive dose of [14C] radiolabelled SHR4640 recovered in urine, faeces and in total, up to Day 10 (approx).
Quantitive analysis of the concentrations of SHR4640 in plasma using the validated LC-MS/MS to obtain pharmacokinetic data. | Up to 10 days (approx) from the start of administration.
  The concentrations of SHR4640 in plasma up to Day 10.
Identification of the main metabolite and biotransformation pathway of SHR4640 and investigation of metabolite in plasma by LC-HR MS. | Up to 10 days (approx) from the start of administration.
  Proportion of different metabolites.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events. | Up to 10 days (approx) from the start of administration.
  Laboratory indicators, 12-lead electrocardiogram (ECG), physical examination,vital signs, adverse events (NCI-CTC AE 5.0), etc.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Soochow University, Suzhou, Jiangsu, China